CLINICAL TRIAL: NCT05037409
Title: A PHASE 1, RANDOMIZED, DOUBLE BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, IMMUNOGENICITY AND PHARMACOKINETICS FOLLOWING SINGLE INTRAVENOUS DOSE OF PF-06823859 IN JAPANESE HEALTHY PARTICIPANTS
Brief Title: Investigation of Safety, Tolerability, Immunogenicity and Pharmacokinetics of Single-Dose of PF-06823859 in Japanese Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: C0251005
Record Dates: First submitted 2021-08-11; First posted 2021-09-08 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PF-06823859 low (Experimental): Participants will receive single intravenous infusion.
  Interventions: Drug: PF-06823859
- PF-06823859 high (Experimental): Participants will receive single intravenous infusion.
  Interventions: Drug: PF-06823859
- Placebo (Placebo Comparator): Participants will receive single intravenous infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-06823859 — low dose or high dose intravenous infusion
  Arms: PF-06823859 high; PF-06823859 low
Drug: Placebo — Intravenous infusion
  Arms: Placebo

SUMMARY:
Purpose of the study is to evaluate the safety, tolerability, immunogenicity and pharmacokinetics (PK) of PF-06823859 following a single intravenous dose of PF-06823859 300 and 900 mg in Japanese healthy adult participants.

DETAILED DESCRIPTION:
Approximately 12 participants are planned to be enrolled into the study. The study consists of 2 cohorts, and approximately 5 participants will be randomized to PF-06823859 and approximately 1 participant will be randomized to placebo in each cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants must be 20 to 55 years of age, inclusive, at the time of signing the Informed Consent Document (ICD).
2. Participants must have 4 biologically Japanese grandparents born in Japan.
3. Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and 12 lead electrocardiogram (ECG).
4. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
5. Body Mass Index (BMI) of 17.5 to 25 kg/m2; and a total body weight >50 kg (110 lb).

   Informed Consent:
6. Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the ICD and in this protocol.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
2. History of human immunodeficiency virus (HIV) infection, hepatitis C or syphilis; positive testing for HIV, hepatitis C antibody (HCVAb) or syphilis at screening.
3. Infection with hepatitis b virus (HBV)
4. Clinically significant abnormality, including but not limited to current, active tuberculosis (TB) or previous inactive TB, general infections, heart failure or malignancy, on chest X ray performed at screening or within 12 weeks of screening.
5. History of autoimmune disorders.
6. History of allergic or anaphylactic reaction to a therapeutic drug or any components in the study intervention.
7. Participants with clinically significant infections, based on which the investigator judges that the participant should not be enrolled in the study, within 28 days prior to the screening visit.
8. Participants with a fever, based on which the investigator judges that the participant should not be enrolled in the study, within the last 7 days prior to dosing.
9. Participants who have evidence of tuberculosis infection.

   * Participants who have been treated or are currently being treated for active or latent tuberculosis infection are to be excluded.
   * Participants with a history of either untreated or inadequately treated latent or active tuberculosis infection are to be excluded.
10. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality or other conditions or situations related to COVID-19 pandemic (eg, Contact with positive case, residence, or travel to an area with high incidence) that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
11. Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.
12. Recent exposure to any live or attenuated live virus vaccines within 6 weeks of admission to central research unit (CRU)

    * The use of COVID-19 vaccines (except for live or attenuated live virus vaccines) are allowed before 14 days prior to Day 1 or after discharge from CRU.
13. Participants who have received PF-0 6823859 or any other interferon (IFN) alpha-or IFN-beta therapy at any time in the past.
14. Previous administration with an investigational drug within 4 months (180 days for biologics) or 5 half lives preceding the first dose of study intervention used in this study (whichever is longer).
15. A positive urine drug test.
16. Screening supine blood pressure (BP) ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥140 mm Hg (systolic) or ≥90 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
17. Screening pulse rate (PR) >100 bpm. If the PR is greater than 100 beat per minute (bpm), the PR should be repeated 2 more times and the average of the 3 PR values should be used to determine the participant's eligibility.
18. Baseline standard 12 lead ECG that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results.
19. Participants with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat test, if deemed necessary:

    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT)level ≥1.5 × upper limit of normal (ULN);
    * Total bilirubin level ≥1.5 × ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
20. A positive COVID-19 test by polymerase chain reaction (PCR) at screening.
21. History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of screening.
22. Blood donation (excluding plasma donations) of approximately ≥400 mL within 3 months or ≥200 mL within a month prior to dosing. Additionally, approximately ≥400 mL within 4 months for female participants.
23. History of sensitivity to heparin or heparin induced thrombocytopenia only if heparin is planned to flush intravenous catheters.
24. History of substance abuse within 12 months of the screening visit.
25. Pregnant females; breastfeeding females.
26. Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
27. Investigator site staff or Pfizer employees directly involved in the conduct of the study, site staff otherwise supervised by the investigator, and their respective family members.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Medical Corporation Shinanokai Shinanozaka Clinic, Shinjuku-ku, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0251005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 13 participants were enrolled and randomized in the study.
Groups:
- Cohort 1: PF-06823859 300 mg: Participants were randomized and administered a single dose of PF-06823859 300 milligrams (mg) as 60 minute intravenous (IV) infusion using a calibrated infusion pump on Day 1 of Cohort 1. Participants were followed up to Day 157.
- Cohort 2: PF-06823859 900 mg: Participants were randomized and administered a single dose of PF-06823859 900 mg as 60 minute IV infusion using a calibrated infusion pump on Day 1 of Cohort 2. Participants were followed up to Day 157.
- Placebo: Participants who were randomized and administered placebo as 60 minute IV infusion using a calibrated infusion pump on Day 1 of each Cohort 1 and Cohort 2 respectively were included in this reporting arm. Participants were followed up to Day 157 (relative to Day 1 of each Cohort).
Period: Blinded Treatment (1 Day)
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Started | 5 | 6 | 2
Treated | 5 | 5 | 2
Completed | 5 | 5 | 2
Not Completed | 0 | 1 | 0
Not completed — Failure to comply with site instruction | 0 | 1 | 0
Period: Follow-up ( Up to Day 157)
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Started | 5 | 5 | 2
Completed | 5 | 5 | 2
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Groups:
- Cohort 1: PF-06823859 300 mg: Participants were randomized and administered a single dose of PF-06823859 300 mg as 60 minute IV infusion using a calibrated infusion pump on Day 1 of Cohort 1. Participants were followed up to Day 157.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 2 | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.80 (14.24) | 33.80 (13.95) | 35.50 (13.44) | 36.17 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 4 | 4 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. SAE was any untoward medical occurrence that at any dose resulted in any of following outcomes/deemed significant for any other reason: death; initial /prolonged inpatient hospitalization; life-threatening; persistent or significant disability/incapacity; congenital anomaly/birth defect and suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic. TEAEs were the events between first dose of study drug and up to Day 157, that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious (if occurred) and all non-serious adverse events.
Time Frame: Day 1 up to maximum of Day 157
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants
  TEAEs | 4 | 1 | 0
  SAEs | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Infusion Related Reaction (IRR)
Description: IRR included AEs potentially related to infusion related reaction and was determined by blind medical review prior to the database release.
Time Frame: Day 1 up to maximum of Day 157
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Infusion Site Reaction
Description: Participants were monitored from start of study intervention infusion until the end of infusion to assess the infusion sites for erythema, induration, ecchymosis, pain, and pruritus, or other observed characteristics after study intervention.
Time Frame: From start of study intervention infusion up to 60 minutes on Day 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Viral Infection
Time Frame: Day 1 up to maximum of Day 157
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants | 0 | 1 | 0

5. Primary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory test abnormalities included hematology: basophils/leukocytes greater than (>)1.2* upper limit of normal (ULN), eosinophils/leukocytes >1.2* ULN, monocytes/leukocytes >1.2* ULN; clinical chemistry: bilirubin > 1.5* ULN, aspartate aminotransferase >3.0* ULN, urate >1.2* ULN; urinalysis: ketones greater than or equal to (>=)1, urine hemoglobin >=1.
Time Frame: Day 1 up to maximum of Day 157
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants | 2 | 4 | 1

6. Primary Outcome: Number of Participants With Vital Sign Abnormalities of Pre-defined Criteria
Description: Vital sign abnormalities were categorized as: a) supine systolic blood pressure: minimum: less than (<) 90 millimeter of mercury (mmHg), maximum decrease from baseline: greater than or equal to (>=) 30 mmHg, maximum increase from baseline: >=30 mmHg; b) supine diastolic blood pressure: minimum: <50 mmHg, maximum decrease from baseline: >=20 mmHg, maximum increase from baseline: >=20 mmHg; c) supine pulse rate: minimum <40 beats per minute (bpm), maximum >120 bpm. Number of participants with any vital sign abnormality were reported in this outcome measure.
Time Frame: From baseline (pre-dose measurement at Day 1) up to Day 157
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities of Pre-defined Criteria
Description: Criteria for ECG abnormalities: maximum PR interval >=300 milliseconds (msec); maximum increase in PR interval from baseline >=25 percent (%) for baseline value of >200 msec; maximum increase in PR interval from baseline >=50% for baseline value of less than or equal to (<=) 200 msec; maximum QRS interval >=140 msec and maximum increase from baseline >=50%; QT interval of >=500 msec; QTcF interval (Fridericia's Correction of QTc interval) mild: >=450 msec to <480 msec, moderate: >=480 msec to <500 msec; increase from baseline >=30 msec to <60 msec and severe: >=500 msec; increase from baseline >=60 msec.
Time Frame: From baseline (pre-dose measurement at Day 1) up to Day 157
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
Number analyzed (Participants) | 5 | 5 | 2
Participants | 0 | 0 | 0

8. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of PF-06823859
Description: Cmax was defined as the maximum observed serum concentration of PF-06823859. Cmax was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: Pre dose on Day 1; 1, 2, 6, 12, 24, 48 and 96 hours post-dose on Day 1; Anytime during site visit at Day 15, 29, 43, 57, 71, 99, 127, 157
Population: Pharmacokinetic (PK) parameter set included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and who had at least 1 of the PK parameters of PF-06823859 of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram per milliliter | 134.4 (16) | 350.1 (10)

9. Secondary Outcome: Dose Normalized Cmax (Cmax [dn]) of PF-06823859
Description: Cmax was maximum observed serum concentration. Cmax (dn) was calculated as Cmax/dose. Cmax (dn) was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: PK parameter set included all participants randomly assigned to study intervention who received at least 1 dose of study intervention and who had at least 1 of the PK parameters of PF-06823859 of interest calculated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter per milligram
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram per milliliter per milligram | 0.4483 (16) | 0.3890 (10)

10. Secondary Outcome: Time to Reach Maximum Observed Serum Concentration (Tmax) of PF-06823859
Description: Tmax was defined as the time to reach maximum observed serum concentration of PF-06823859 and was observed directly from data. Tmax was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Hours | 2.000 [1.00 to 6.00] | 2.000 [1.00 to 2.00]

11. Secondary Outcome: Area Under the Curve From Time Zero Extrapolated to Infinite Time (AUCinf) of PF-06823859
Description: AUCinf was calculated as AUClast + (Clast*/kel), where Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel = terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. Area under the curve from time zero to last quantifiable concentration (AUClast) was determined using the linear/log trapezoidal rule. AUCinf was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram*hour per milliliter | 68070 (12) | 178000 (16)

12. Secondary Outcome: Dose Normalized AUCinf (AUCinf [dn]) of PF-06823859
Description: AUCinf (dn) was calculated as AUCinf/dose. Where AUCinf was calculated as AUClast + (Clast*/kel), where Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel = terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUClast was determined using the linear/log trapezoidal rule. AUCinf [dn] was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour/milliliter/milligram
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram*hour/milliliter/milligram | 227.1 (12) | 197.8 (16)

13. Secondary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of PF-06823859
Description: AUClast was determined using the linear/log trapezoidal rule. AUClast was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram*hour per milliliter | 66120 (12) | 173000 (14)

14. Secondary Outcome: Dose Normalized AUClast (AUClast [dn]) of PF-06823859
Description: AUClast(dn) was calculated as AUClast/dose. AUClast(dn) was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour/milliliter/milligram
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram*hour/milliliter/milligram | 220.4 (12) | 192.2 (14)

15. Secondary Outcome: Area Under the Curve From Time Zero to 14 Days (336 Hours) Post-Dose (AUC14day) of PF-06823859
Description: AUC14day = area under the serum concentration-time profile from time 0 to 14 days post-dose. AUC14day was determined using the linear/log trapezoidal rule. AUC14day was analyzed and reported consolidated for all the time-points through Day 1 to Day 14.
Time Frame: Pre dose on Day 1; 1, 2, 6, 12, 24, 48, 96 and 336 hours post dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram*hour per milliliter | 22170 (10) | 61170 (8)

16. Secondary Outcome: Area Under the Curve From Time Zero to 28 Days (672 Hours) Post-Dose (AUC28day) of PF-06823859
Description: AUC28day = area under the serum concentration-time profile from time 0 to 28 days post-dose. AUC28day was determined using the linear/log trapezoidal rule. AUC28day was analyzed and reported consolidated for all the time-points through Day 1 to Day 28.
Time Frame: Pre dose on Day 1; 1, 2, 6, 12, 24, 48, 96, 336 and 672 hours post dose on Day 1
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram*hour per milliliter
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Microgram*hour per milliliter | 35040 (10) | 95250 (10)

17. Secondary Outcome: Terminal Half-Life (t1/2) of PF-06823859
Description: Terminal half-life (t1/2) is the time for the serum concentration of a drug to decrease by half of its initial concentration. T1/2 was determined using loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. T1/2 was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Days | 32.42 (0.70852) | 31.42 (4.9505)

18. Secondary Outcome: Systemic Clearance (CL) of PF-06823859
Description: CL was calculated as Dose divided by AUCinf. AUCinf was calculated as AUClast + (Clast*/kel), where Clast* was the predicted serum concentration at the last quantifiable time point estimated from the log-linear regression analysis and kel = terminal phase rate constant calculated by a linear regression of the log-linear concentration-time curve. AUClast was determined using the linear/log trapezoidal rule. CL was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Liter per hour | 0.004406 (12) | 0.005061 (16)

19. Secondary Outcome: Steady-State Volume of Distribution (Vss) of PF-06823859
Description: Volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Vss was calculated as CL*Mean residence time (MRT). MRT was calculated as AUMCinf/AUCinf - DOF/2, where AUMCinf is the area under the moment curve from time 0 extrapolated to infinity and DOF is the duration of the IV infusion. Vss was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Liter | 4.304 (10) | 4.737 (7)

20. Secondary Outcome: Mean Residence Time (MRT) of PF-06823859
Description: MRT was calculated as AUMCinf/AUCinf - DOF/2, where AUMCinf is the area under the moment curve from time 0 extrapolated to infinity and DOF is the duration of the IV infusion. MRT was analyzed and reported consolidated for all the time-points through Day 1 to Day 157.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Days | 40.69 (8) | 38.99 (15)

21. Secondary Outcome: Number of Participants With Positive Anti-Drug Antibody (ADA) and Neutralizing Antibodies (NAb) for PF-06823859
Description: A participant was ADA positive if (1) baseline ADA titer was missing or negative and participant had >= 1 post-treatment positive titer (treatment-induced), or (2) positive ADA titer at baseline and had a >= 0.602 unit increase in titer from baseline in >= 1 post-treatment sample (treatment-boosted). A participant was NAb positive, if baseline was missing or negative and participant had >= 1 post-treatment positive. NAb-negative participants included participants who were ADA negative or ADA-positive participants tested post-treatment negative in the NAb assay. Participants who were NAb positive at baseline and had >= 1 post-treatment positive were handled as NAb negative.
Time Frame: Day 1 maximum up to Day 157
Population: Immunogenicity analysis set included all participants randomly assigned to study intervention who received at least 1 dose of study intervention with at least 1 post-treatment anti-drug (PF-06823859) antibody determination. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg
Number analyzed (Participants) | 5 | 5
Participants
  Positive ADA | 1 | 1
  Positive NAb | 1 | 1

ADVERSE EVENTS:
Time Frame: Day 1 up to maximum of Day 157
Description: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Arm/Group | Cohort 1: PF-06823859 300 mg | Cohort 2: PF-06823859 900 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 4/5 | 1/5 | 0/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: PF-06823859 300 mg (N=5) | Cohort 2: PF-06823859 900 mg (N=5) | Placebo (N=2)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0
Vaccination site pain (General disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT05037409/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-14): https://cdn.clinicaltrials.gov/large-docs/09/NCT05037409/SAP_001.pdf